CLINICAL TRIAL: NCT00746161
Title: A Prospective Randomized Controlled Trial Comparing Double Tract Method With Roux-en-Y Method After Total Gastrectomy in Patients With Gastric Cancer
Brief Title: Evaluation of Double Tract Reconstruction After Total Gastrectomy in Patients With Gastric Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wakayama Medical University (Other)
Responsible Party: Second Department of Surgery, Wakayama Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WMU-GC02
Record Dates: First submitted 2008-09-02; First posted 2008-09-03 (Estimated); Last update posted 2008-09-04 (Estimated); Status verified 2008-09

CONDITIONS: Gastric Cancer
Keywords: total gastrectomy; double tract reconstruction; gastric cancer; Total gastrectomy in patients with gastric cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Roux-en-Y
  Interventions: Procedure: Reconstruction after total gastrectomy
- 2 (Experimental): double tract reconstruction
  Interventions: Procedure: Reconstruction after total gastrectomy

INTERVENTIONS:
Procedure: Reconstruction after total gastrectomy — Roux-en-Y
  Arms: 1
Procedure: Reconstruction after total gastrectomy — double tract reconstruction
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the double tract reconstruction after total gastrectomy in patients with gastric cancer. A prospective randomized controlled trial was conducted to compare double tract method with Roux-en-Y method

DETAILED DESCRIPTION:
Patients with gastric cancer were intraoperatively randomized for R-Y reconstruction or DT reconstruction after total gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven adenocarcinoma without esophageal invasion, tumor status T1-2
* Age 80 years or younger
* No distant metastasis

Exclusion Criteria:

* Carcinoma in the remnant stomach
* Stage intravenous (IV)
* History of laparotomy
* History of serious heart disease
* Liver cirrhosis or chronic liver disease with indocyanine green excretion test at 15 min of 15% or more
* Absence of informed consent

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2002-04; Primary Completion 2008-01 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
The %body weight ratio | 12 months after operation

SECONDARY OUTCOMES:
preoperative complication, PNI and QOL score | within one month, and 3 and 12months after operation

CONTACTS AND LOCATIONS:
Overall Officials: Makoto Iwahashi, Principal Investigator — Second Department of Surgery, Wakayama Medical University
Locations (1):
- Second Department of Surgery, Wakayama Medical University, Wakayama, Wakayama, Japan

REFERENCES:
- [Derived] Iwahashi M, Nakamori M, Nakamura M, Naka T, Ojima T, Iida T, Katsuda M, Ueda K, Yamaue H. Evaluation of double tract reconstruction after total gastrectomy in patients with gastric cancer: prospective randomized controlled trial. World J Surg. 2009 Sep;33(9):1882-8. doi: 10.1007/s00268-009-0109-0. PMID 19548028